CLINICAL TRIAL: NCT07177118
Title: A Prospective, Open-Label, Randomized Controlled Study of Risankizumab (an IL-23 Inhibitor) for the Treatment of Fibrostenotic Crohn's Disease
Brief Title: Risankizumab for Fibrostenotic Crohn's Disease Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Taizhou Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Fang Wu, Chief Physician, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Risankizumab
Record Dates: First submitted 2025-09-05; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease; Crohn Disease and Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Ustekinumab; risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ustekinumab (Active Comparator): Ustekinumab group (induction phase with intravenous equivalent doses at weeks 0 and 8, maintenance phase with 90 mg subcutaneously every 8 weeks)
  Interventions: Drug: Ustekinumab
- risankizumab (Experimental): Risankizumab group (induction phase with intravenous 600 mg at weeks 0, 4, and 8, maintenance phase with 360 mg subcutaneously every 8 weeks)
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab group (induction phase with intravenous equivalent doses at weeks 0 and 8, maintenance phase with 90 mg subcutaneously every 8 weeks)
  Arms: ustekinumab
Drug: Risankizumab — Risankizumab group (induction phase with intravenous 600 mg at weeks 0, 4, and 8, maintenance phase with 360 mg subcutaneously every 8 weeks)
  Arms: risankizumab

SUMMARY:
This study, titled "IL-23 Inhibitor Ustekinumab for the Treatment of Fibrotic Crohn's Disease: A Prospective, Open-Label, Randomized Controlled Study," is conducted by researchers from the First Affiliated Hospital of Wenzhou Medical University. The primary aim of this research is to evaluate the efficacy and safety of ustekinumab, an IL-23 inhibitor, for patients with fibrostenotic Crohn's disease (CD) who have failed standard treatments.

The study is a prospective, open-label, randomized controlled trial involving 260 participants across three major hospitals: the First Affiliated Hospital of Wenzhou Medical University, Taizhou Hospital of Zhejiang Province, and the Second Affiliated Hospital of Wenzhou Medical University. The participants are divided into two groups: one receiving ustekinumab and the other receiving a placebo. The study is designed to assess whether ustekinumab can improve clinical outcomes and reduce fibrosis progression in patients with fibrotic CD.

The study involves a comprehensive assessment of participants, including clinical history, physical examination, laboratory tests, and imaging studies. Key inclusion criteria include age between 18-80 years, confirmed diagnosis of fibrostenic CD, and failure of conventional or biological therapies. Participants are excluded if they are under 18, pregnant, breastfeeding, or have certain medical conditions that could interfere with the study.

The primary endpoint of the study is a clinical-imaging composite endpoint, which includes imaging assessment of bowel wall thickness and clinical symptoms. Secondary endpoints include safety, tolerability, and various functional and quality of life indicators. The study also explores the potential of ustekinumab to modulate immune responses and fibrosis-related biomarkers.

The study is expected to run from October 2025 to October 2028, with follow-up visits scheduled at regular intervals. The results will provide valuable insights into the potential of ustekinumab as a novel treatment for fibrotic CD, offering a new therapeutic option for patients who do not respond to existing treatments.

This research is crucial because fibrotic CD is a severe and progressive disease with limited treatment options. Ustekinumab, by targeting the IL-23 pathway, may offer a more effective and targeted approach to manage this condition. The study's findings could significantly impact clinical practice and improve patient outcomes.

For more detailed information, please refer to the study protocol document titled "IL-23 Inhibitor Ustekinumab for the Treatment of Fibrotic Crohn's Disease: A Prospective, Open-Label, Randomized Controlled Study" dated September 2, 2025. For further inquiries, contact the principal investigators Dr. Wu Fang or Dr. Wu Xiaoli at the First Affiliated Hospital of Wenzhou Medical University.

DETAILED DESCRIPTION:
Summary of the plan

Project Name: Prospective, Open-label, Randomized Controlled Study on the Treatment of Fibrostenosing Crohn's Disease with IL-23 Inhibitor Ruxolitinib

Research purpose Main purpose:

Evaluate the effectiveness of full-course (induction + maintenance) treatment with Lentilisinib in participants with fibrosing Crohn's disease who have failed standard therapy

Secondary objectives:

Evaluate the safety and tolerability of participants in the study of fibrosing Crohn's disease who have failed standard treatment after receiving the full course (induction + maintenance) of Lentilimab, and further observe the preliminary efficacy (radiographic remission rate, clinical response rate, surgery-free survival rate, progression-free survival, and reported outcomes, etc.) Study Subjects: The study subjects are research participants aged between 18 and 80 years, of either gender, with endoscopically and histologically confirmed fibrosing Crohn's disease. These participants have either failed standard treatment or have contraindications/intolerances, and plan to receive treatment with lecanicizumab or ustanumab for the first time. During the screening phase, all study participants must confirm through medical history inquiry and medical record review that they have never used lecanicizumab or ustanumab. If they have used other biologics, they must complete a preset washout period (those who have used any TNF-α monoclonal antibody must discontinue for ≥8 weeks) to ensure that the effects of previous medications have been eliminated. Study participants who have already begun treatment with lecanicizumab or ustanumab will not be included to avoid disrupting randomization, confounding baseline assessments, interfering with safety signals, and violating ethical fairness.

Sample size: 130 cases in each group, totaling 260 individuals Inclusion criteria: ① Age range of 18-80 years, with no gender restrictions

* Voluntarily sign the informed consent form

  ③ Endoscopic and histological confirmation of fibrosclerosing Crohn's disease, and meeting the following criteria:
  * Symptoms suggestive of fibrostenosis, such as spasms, dietary restrictions or changes, postprandial vomiting, and abdominal pain;
  * Endoscopy or imaging confirms new-onset fibrotic stenosis (not caused by previous dilation/stenting);
  * The length of the stenosis is less than 10 cm, and there are a maximum of 2 stenoses in a single intestinal segment;

    * Clinical manifestations of intestinal obstruction or sub-obstruction ⑤ Previous insufficient efficacy, intolerance, or contraindications to conventional or biological agents (such as azathioprine, 6-mercaptopurine, methotrexate, TNF-α monoclonal antibody, etc.) ⑥ Plan to receive treatment with lecaniclib or ustunumab for the first time ⑦ Have not previously used risankizumab or ustekinumab; if other biologics have been used, they have been discontinued for ≥ the specified washout period (TNF-α monoclonal antibody ≥ 8 weeks) Exclusion criteria: ① Age <18 or >80 years old
* Refusal or inability to sign the informed consent form

  * No symptoms of Crohn's disease such as spasm, dietary restrictions or changes, vomiting after eating, and abdominal pain

    * Stenosis has undergone stenting and/or dilation treatment (<1 year)

      * Pregnancy, lactation, or preparation for pregnancy

        * Endoscopy is not feasible or there are clinical conditions incompatible with endoscopy

          * Combined with abscess, fistula, or active complex stenosis (not limited to the stenotic segment) ⑧ The length of the stenosis is ≥10 cm or the number of stenoses is >2

            ⑨ Severe coagulation dysfunction (platelet count < 50,000; INR > 1.5)

            ⑩ Patients with end-organ failure, HIV-positive, uncontrolled infection, or a history of malignancy within the past 5 years

            ⑪ Has received or started treatment with durvalumab or ustekinumab

            ⑫ The researcher judges that there are other situations that make the participant unsuitable for participating in this clinical study Trial Design: This study is a multicenter, open-label, randomized, controlled trial. It intends to enroll 260 participants with fibrosing stricturing Crohn's disease who have failed standard treatment. Participants will be randomly assigned in a 1:1 ratio to the ustekinumab group (equivalent intravenous doses at weeks 0 and 8 during the induction phase, and 90 mg subcutaneously every 8 weeks during the maintenance phase) or the lecaniclib group (600 mg intravenously at weeks 0, 4, and 8 during the induction phase, and 360 mg subcutaneously every 8 weeks during the maintenance phase). The treatment duration is 52 weeks, followed by a 24-week follow-up period (approximately 6 months) after the last dose. The primary endpoint is the achievement rate of the clinical-radiological composite endpoint, which includes: 1. No radiological progression of strictures: Changes in the length or diameter of intestinal strictures assessed by MR/CTE compared to baseline are less than 20%; 2. Survival without clinical obstruction events: No intestinal obstruction requiring hospitalization or surgical/endoscopic intervention occurs. Secondary endpoints include safety (TEAEs, SAEs), radiological remission rate, clinical response rate, surgery-free survival rate, progression-free survival period, reported outcomes, etc. Biomarkers such as peripheral blood IL-23 and TIMP-1 will be dynamically monitored to explore predictive factors for efficacy.

Endpoint indicators: Primary endpoint:

Clinical-radiological composite endpoint, meeting all of the following criteria -

1. No progression of stenosis on imaging: The change in the length or diameter of intestinal stenosis as assessed by MR/CTE compared to baseline is less than 20%
2. Survival without clinical obstruction events: No intestinal obstruction requiring hospitalization or surgical/endoscopic intervention

Secondary endpoints:

1. Drug safety

   * Incidence of treatment-emergent adverse events (TEAEs) during treatment (including infusion reactions, infections, liver dysfunction, etc.)
   * Incidence of serious adverse events (SAEs) and adverse events leading to drug discontinuation (intestinal obstruction, perforation, severe infection, etc.) The incidence of abnormalities in vital signs, electrocardiogram, physical examination, laboratory tests, and changes compared to baseline
2. Drug efficacy 2.1 Objective remission indicators

   * Imaging response rate (MR/CTE assessment of intestinal wall thickness reduction ≥25%)
   * Clinical response rate (CDAI decrease ≥100 points or clinical remission) 2.2 Disease control indicators
   * Surgery-free survival rate (the proportion of patients who are free from intestinal resection or stricture plasty at 1 year/2 years)
   * Progression-free survival (PFS) 2.3 Functional improvement indicators Patient-Reported Outcomes (PROs): Improvement in Obstructive Symptom Score (OSS) ≥50%; Increase in IBD-Q Quality of Life Score ≥20 points

Exploratory endpoint:

Dynamic changes of serum/tissue fibrosis markers (TIMP-1, COL3A1, TGF-β)

* Imaging elasticity assessment (ultrasound/MR elastography) of intestinal wall fibrosis degree changes
* Gut microbiota profile and peripheral blood levels of cytokines related to the IL-23/IL-17 pathway Statistical analysis was conducted using SAS 9.4 (or later) software. Continuous variables are described using mean, standard deviation, median, minimum, and maximum values, while count and ordinal data are described using frequency and percentage.

The statistical analysis sets involved in this study are as follows:

Full Analysis Set (FAS): all study participants who were enrolled and received at least one treatment.

Safety Set (SS): individuals who have received at least one treatment and have post-treatment safety indicators The recorded research participants. Distribution of study participants Based on the description of the screened population, the screening and enrollment status of study participants will be summarized. For study participants who failed to be screened, the reasons for their failure will be summarized. Based on the enrolled population, the enrollment status and trial completion status of each dose group will be summarized. For study participants who withdrew from the study, the reasons for their withdrawal will be summarized.

Demographic data and baseline analysis FAS will be used for demographic analysis. The characteristics of study participants include baseline medical history and disease characteristics. Statistical descriptions will be provided for the demographic and baseline characteristics of study participants across different dosage groups, categorized by variable type.

Study on product exposure and analysis of concomitant medication/treatment Conduct analysis based on SS. Descriptive statistics of cell infusion frequency, dosage, and infusion duration.

Previous medications and concomitant medications were encoded using the WHO DRUG dictionary, summarized based on the second-level classification of ATC and PT, and the number of cases and proportions were calculated.

List a detailed inventory of previous medications/treatments and concurrent medications/treatments.

Effectiveness analysis Conduct analysis based on FAS. To calculate the stenosis-free progression rate, the Clopper-Pearson method was used to compute its 95% confidence interval (CI).

For survival rate without surgery, imaging response rate, and clinical response rate, the Kaplan-Meier method was used for analysis. The number of events, number of censored cases, and their percentages were listed, and the median time and its 95% confidence interval (CI) were calculated.

Other continuous indicators (changes in intestinal wall thickness, serum fibrosis marker levels) were analyzed using a mixed linear model.

Safety analysis Analyze based on SS. Adverse events are coded according to the ICH Medical Dictionary for Regulatory Activities (MedDRA).

Calculate the incidence of treatment-emergent adverse events (TEAE)/reactions, serious adverse events/reactions, and adverse events/reactions leading to early withdrawal.

Summarize the number of cases and instances of adverse events/reactions, serious adverse events/reactions, and adverse events/reactions leading to early withdrawal during the treatment period according to SOC, PT, and severity, and calculate the incidence rate.

List a detailed list of cases involving various adverse events/reactions, serious adverse events/reactions, and adverse events/reactions leading to early withdrawal.

List the cross-tabulation of laboratory tests, electrocardiogram, and physical examination before and after medication.

Descriptive statistics of laboratory tests, electrocardiogram, changes in vital signs from baseline, and actual measured values.

List a detailed list of abnormal values from laboratory tests, electrocardiogram, and physical examination.

Research period: October 2025 - October 2028

ELIGIBILITY:
Inclusion Criteria:

- Here's the translation of the provided criteria into English:

1. Age between 18 and 80 years old, with no gender restrictions.
2. Voluntarily sign an informed consent form.
3. Diagnosed with fibrostenosing Crohn's disease by endoscopy and histology, and meet the following criteria:

   * Presence of symptoms indicating fibrostenosis, such as cramping, dietary restrictions or changes, postprandial vomiting, and abdominal pain;
   * Endoscopic or radiological confirmation of new fibrotic stenosis (not caused by previous dilation/stenting);
   * The length of stenosis is less than 10 cm, and there are no more than 2 stenoses in a single intestinal segment;
4. Clinical manifestations of intestinal obstruction or sub-obstruction.
5. Insufficient efficacy, intolerance, or contraindications to conventional or biological agents (azathioprine, 6-mercaptopurine, methotrexate, TNF-α inhibitors, etc.).
6. Plan to receive treatment with risankizumab or ustekinumab for the first time.
7. Have not previously used risankizumab or ustekinumab; if other biological agents have been used, they have been discontinued for at least the specified washout period (TNF-α inhibitors ≥8 weeks).

Exclusion Criteria:

* Here is the translation of the exclusion criteria into English:

  1. Age less than 18 or greater than 80 years old.
  2. Refusal or inability to sign the informed consent form.
  3. Absence of symptoms of fibrostenotic Crohn's disease, such as cramping, dietary restrictions or changes, postprandial vomiting, and abdominal pain.
  4. Prior stenting and/or dilation treatment for stenosis (within less than 1 year).
  5. Pregnancy, lactation, or planning to conceive.
  6. Inaccessible endoscopy or presence of clinical conditions incompatible with endoscopy.
  7. Presence of abscesses, fistulas, or active complex strictures (not limited to the strictured segment).
  8. Stenosis length of 10 cm or greater, or more than 2 strictures in a single intestinal segment.
  9. Severe coagulation dysfunction (platelet count < 50,000; INR > 1.5).
  10. Presence of end-stage organ failure, positive for Human Immunodeficiency Virus, uncontrolled infections, or a history of malignant tumors within the past 5 years.
  11. Having received or started treatment with risankizumab or ustekinumab.
  12. Investigator determines other conditions that make participation in this clinical study unsuitable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2028-06-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Radiological Composite Endpoint | up to 24 weeks
  No progression of stenosis: Assessment by MRI/CTE shows a change in the length or diameter of the intestinal stenosis of less than 20% compared to baseline.

IPD SHARING:
Plan to Share IPD: Yes
This study plans to share de-identified individual participant data (IPD) with qualified researchers upon request. The data will include clinical outcomes, demographic information, and treatment responses, excluding any personally identifiable information to ensure participant privacy. Access to the data will be granted through a secure data-sharing platform, and interested researchers will need to submit a research proposal outlining the intended use of the data. The sharing of IPD will be subject to approval by an independent data access committee to ensure that the proposed research aligns with ethical standards and scientific integrity.
Supporting Information: Study Protocol, ICF